CLINICAL TRIAL: NCT06117475
Title: Short-term Outcomes of Posterior Corpectomy in Thoracolumbar Spinal Metastatsis in Assiut University Hospitals
Brief Title: Posterior Corpectomy in Thoracolumbar Spinal Metastatsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Mahmoud Ahmed Mohammed, Assiut lecturer, Assiut University
Other Study IDs: Spinal metastatses
Record Dates: First submitted 2023-10-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Spine Metastases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Posterior corpectomy — Removal of posterior portion of vertebrae by posterior approach

SUMMARY:
To analyze the short-term outcomes of posterior corpectomy of patients with thoracolumbar spinal metastasis in spine unit in Assiut University hospital regarding the pain control , neurological status , complication and ambulatory status as well as mortality rate.

DETAILED DESCRIPTION:
The metastasis is the spread of cancer from one part of the body to another. Two-thirds of patients with cancer will develop bone metastases. Breast, prostate and lung cancer are responsible for more than 80% of cases of metastatic bone disease. A spinal metastasis may cause pain, instability and neurological injuries.

* The spine is the most common site of bone metastasis . It is estimated that over the 10% of patients with cancer will develop a symptomatic spinal metastasis . Algra et al. suggest that the initial anatomic location of metastases within vertebrae is in the posterior portion of the body.
* Spinal metastases are the most common tumors of the spine, comprising approximately 90% of masses encountered with spinal imaging. Within the spinal column, metastasis is more commonly found in the thoracic region, followed by the lumbar region, while the cervical region is the least likely place professionals find metastasis .
* Spinal metastases most commonly affect the vertebral bodies of the spinal column, and spinal cord compression is an indication for surgery. Commonly, an open posterior approach is employed to perform a transpedicular, costotransversectomy or lateral extracavitary corpectomy. Because of the short life expectancies in patients with metastatic spinal disease, decreasing the morbidity of surgical treatment and recovery time is critical.
* At present, both surgical and nonsurgical treatments are used for the treatment of spinal tumors, however, treatment outcome is dependent on various factors, such as patient age, overall health of the patient .
* When treating patients with vertebral metastases, surgical strategy is mainly based on life expectancy, primary site of tumor, and staging. This helps determine which patients will benefit from surgery and the type of procedure. Tokuhashi developed a score to determine life expectancy in order to facilitate the treatment modality decision .
* Vertebral corpectomy refers to the removal of one or more vertebral bodies from the spine, as well as the intervertebral discs above and below the surgical level.

Corpectomies may be accomplished through a multitude of approaches. Posterior approaches have been associated with less intraop- erative blood loss, complications, shorter operative time, and better pul- monary function post-operation compared to anterior approaches .

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years old Patient diagnosed as cancer Intractable pain Progressive neurologic comprise Radioresistant tumors

* Failure of radiotherapy
* Failure of chemotherapy
* Fit for surgery

Exclusion Criteria:

Patient younger 18 years old spinal 1ry tumor

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed as a spinal metastatsis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of patient life postoperatively | 5Q-ED score through complete the study about 1to 1.5 years
  Measure quality of life postoperatively by mobility, self care , usual activity ( e.g work, study, housework ) , pain /discomfort and anxiety and depression by 5Q-ED score ( EUROQOL EUROQOL 5 Dimension 5 levels ). EQ-5D-5L profile data can be summarised in the same way. 11111 again means no problem on any of the five dimensions of health and the worst health state is 55555.
  1 means no problem , 5 means unable to do

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Gamal, Professor, Principal Investigator — Assiut University; Essam Elmorshidy, MD, Principal Investigator — Assiut University

REFERENCES:
- [Background] Maccauro G, Spinelli MS, Mauro S, Perisano C, Graci C, Rosa MA. Physiopathology of spine metastasis. Int J Surg Oncol. 2011;2011:107969. doi: 10.1155/2011/107969. Epub 2011 Aug 10. PMID 22312491
- [Background] Algra PR, Heimans JJ, Valk J, Nauta JJ, Lachniet M, Van Kooten B. Do metastases in vertebrae begin in the body or the pedicles? Imaging study in 45 patients. AJR Am J Roentgenol. 1992 Jun;158(6):1275-9. doi: 10.2214/ajr.158.6.1590123.
- [Background] Mundy GR. Metastasis to bone: causes, consequences and therapeutic opportunities. Nat Rev Cancer. 2002 Aug;2(8):584-93. doi: 10.1038/nrc867. PMID 12154351
- [Background] Lau D, Chou D. Posterior thoracic corpectomy with cage reconstruction for metastatic spinal tumors: comparing the mini-open approach to the open approach. J Neurosurg Spine. 2015 Aug;23(2):217-27. doi: 10.3171/2014.12.SPINE14543. Epub 2015 May 1. PMID 25932599
- [Background] Bilsky MH, Lis E, Raizer J, Lee H, Boland P. The diagnosis and treatment of metastatic spinal tumor. Oncologist. 1999;4(6):459-69. PMID 10631690
- [Background] Gruenberg M, Mereles ME, Willhuber GOC, Valacco M, Petracchi MG, Sola CA. Usefulness of Tokuhashi Score in Survival Prediction of Patients Operated for Vertebral Metastatic Disease. Global Spine J. 2017 May;7(3):260-265. doi: 10.1177/2192568217699186. Epub 2017 Apr 11. PMID 28660109
- [Background] Lin B, Chen ZW, Guo ZM, Liu H, Yi ZK. Anterior Approach Versus Posterior Approach With Subtotal Corpectomy, Decompression, and Reconstruction of Spine in the Treatment of Thoracolumbar Burst Fractures: A Prospective Randomized Controlled Study. J Spinal Disord Tech. 2012 Aug;25(6):309-317. doi: 10.1097/BSD.0b013e3182204c53. PMID 21637134